CLINICAL TRIAL: NCT06573879
Title: Effect of Eccentric Exercise on Musculus Triceps Surae Muscle Architecture, Muscle Strength, and Performance in Young Volleyball Players
Brief Title: Effect of Eccentric Exercise on Musculus Triceps Surae Muscle Architecture, Muscle Strength, and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Seda GÖZENER CANBÜLBÜL, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-7779
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Muscle Architecture
Keywords: Muscle architecture; Muscle strength; Jumping performance

STUDY DESIGN:
Intervention Model Description: The study participants will be divided into two different groups - a control group and an exercise group.
  Control Group: 15 Exercise Group: 15 Exercise Program: A strength training program will be provided to the exercise group, carried out 3 days a week with 3 sets of 10 repetitions each day.
  Total Duration: 8 Weeks (approximately 2 months)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Group (EG) (Experimental): Exercise Group (EG) is the first arm of the study in which volleyball athlete participants performed eccentric exercises in addition to their exercise routines.
  Interventions: Behavioral: Eccentric Exercise
- Control Group (CG) (No Intervention): Control Group (CG) is the second arm of the study, where volleyball athletes only continued their exercise routines and no external intervention was made.

INTERVENTIONS:
Behavioral: Eccentric Exercise — It was investigated whether volleyball athlete participants would develop muscle architecture, muscle strength and performance parameters differently from the control group by performing eccentric exercises in addition to their exercise routines.
  Arms: Exercise Group (EG)

SUMMARY:
This study investigates the architecture, muscle strength, and performance of skeletal muscles. Skeletal muscles constitute a mass of muscle fascicles connected to bones via tendons. Muscle architecture is defined as the geometric arrangement of muscle fiber bundles in relation to the axis that generates force. This arrangement influences the muscle's contraction speed, force generation capacity, and range of motion. Ultrasonography is a method for examining muscle morphology without radiation exposure. The architectural features of muscles have been a proven method for evaluating and enhancing muscle function. The purpose of this study is to examine the effects of eight weeks of eccentric exercises on the right and left triceps surae muscles in young volleyball players. This investigation aims to contribute to the literature concerning muscle architecture. The study will be conducted using statistical analysis and the SPSS program.

The study has obtained ethical approval and will be conducted at Istanbul Medipol University. Thirty healthy young volleyball players will be involved in this research. The participants' muscle architecture, strength, and performance will be measured. Additionally, the impact of eccentric exercises will be examined, and statistical data analysis will be carried out.

Ultimately, this study aims to explore the effects of eccentric exercise on the muscle architecture and performance of young volleyball players, aiming to contribute to the literature by understanding and enhancing muscle function and performance.

DETAILED DESCRIPTION:
Skeletal muscles are organized masses of muscle fascicles covered with connective tissue, attached to bones at both ends through tendons. The volume of a muscle is largely determined by the total number of sarcomeres within that muscle. Sarcomeres are approximately 1 µm in diameter and 2-3 µm in length. These functional units are aligned end-to-end to form myofibrils, which are packed parallel to create muscle fibers (approximately 50 µm in diameter in humans). Bundling these muscle fibers in parallel forms fascicles (approximately 1 to 3 mm in diameter in humans), which, in turn, combine in parallel to create muscles.

Muscle architecture is defined as the geometric arrangement of muscle fiber bundles concerning the axis that generates force. Muscles with fibers extending longitudinally along the muscle length possess longitudinal muscle architecture, while muscles with fibers running at a certain angle along the muscle length and containing shorter fibers possess pennate or multipennate muscle architecture.

This arrangement affects a muscle's contraction speed, force generation capacity, and range of motion known as 'excursion'. In pennate muscles, bundles of fibers, referred to as fascicles, are positioned obliquely and attach to the muscle's aponeuroses. The angle at which a fascicle attaches to the aponeurosis defines the pennation angle. The distance between epimysiums (superficial and deep aponeuroses in ultrasonography) defines the anatomical muscle thickness. These parameters of skeletal muscle architecture are measured through muscle physiology and biomechanical studies to determine the anatomical and contractile characteristics of the muscles. Typical parameters included in architectural analysis are fiber length, pennation angle, and physiological cross-sectional area.

Ultrasonography enables the examination of muscle morphology without radiation exposure. Fascicle length, pennation angle, and muscle thickness can be measured in vivo using two-dimensional (2D) B-mode ultrasonography. In ultrasonographic imaging, normal muscle tissue appears as a structure with low echo intensity. As the epimysium surrounding the muscle is quite reflective, the muscle's boundaries are clearly visible.

While skeletal muscles show significant structural similarities at a microscopic level, muscle architecture is the fundamental factor creating differences in strength and functional capabilities. Understanding the architectural features of muscles allows for the effective assessment and improvement of muscle function. Loading placed on muscles results in an adaptive process leading to muscle development. Muscle architecture allows the macroscopic understanding and interpretation of this adaptation process.

Although muscle strength is primarily determined by genetic structure, it is also influenced by factors such as the level of physical activity, age, gender, motivation, and nutrition. The magnitude of the cross-sectional area of a muscle - which includes the number of engaged fibrils and the size of these fibrils - accounts for the muscle's strength. Developing these aspects is achievable through exercise.

Exercise is defined as a planned, structured, intentional, and continuous activity aimed at enhancing physical fitness. Strength training exercises are designed to increase muscle strength and endurance by applying resistance.

One type of exercise, eccentric exercises, involves movements against gravity using body weight or additional loads. Eccentric exercises are utilized to increase muscle strength and mass. More muscle strength can be generated through these exercises compared to concentric or isometric exercises. Due to their features in injury prevention, rehabilitation, and improving physical fitness in healthy individuals, eccentric training has become quite popular. However, findings regarding the effects of eccentric training on the m. triceps surae are contradictory. Some studies show that eccentric training promotes an increase in muscle fiber length, pennation angle, and muscle thickness, while others find no changes in these architectural outcomes. This might be due to the non-uniform distribution of loads among synergistic muscles and the observation of different mechanical loads for different components of the m. triceps surae. Additionally, short muscle fibers are more sensitive to muscle damage caused by eccentric training compared to long muscle fibers. Considering the differences in architectural features of m. triceps surae segments (GM, GL, SO, and PL), eccentric exercises may produce different results.

The aim of the study is to investigate the effects of 8 weeks of eccentric exercises, performed three times a week for a total of 24 sessions, on the muscle architecture of the m. triceps surae in healthy female participants. Ultrasonography will be utilized to measure fascicle length, pennation angle, and muscle thickness in the gastrocnemius medialis (GM), gastrocnemius lateralis (GL), soleus (SO), and plantaris (PL) muscles before and after the exercise program. It is hypothesized that an 8-week eccentric exercise program will increase fascicle length, pennation angle, and muscle thickness in the m. triceps surae muscles. The architectural adaptations to eccentric exercises must be understood to develop effective exercise programs for improving muscle strength and function.

ELIGIBILITY:
Inclusion Criteria:

* Having healthy lower extremities
* Being a volleyball athlete for at least the last 5 years
* Full range of motion in the lower extremity

Exclusion Criteria:

* Systemic inflammatory joint disease for both groups
* Having had an acute or chronic lower extremity injury during the last 6 months
* Having any orthopedic disorder in the lower extremity
* Severe pain or limitation of movement in the lower extremity
* Previous lower extremity surgery
* Participant noncompliance during testing
* Presence of severe effusion and severe limitation in joint movement

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Muscle Architecture- muscle thickness | 5 months
  Muscle architecture of the gastrocnemius medialis, lateralis, and soleus muscles are visualized by the USG device.
  Their muscle thickness (mm) is measured and recorded.
Muscle Architecture- fiber length | 5 months
  Muscle architecture of the gastrocnemius medialis, lateralis and soleus muscles are visualized by the USG device.
  Their fiber length (mm) is measured and recorded.
Muscle Architecture- pennation angle (degree) | 5 months
  Muscle architecture of the gastrocnemius medialis, lateralis and soleus muscles are visualized by the USG device.
  Their pennation angle (degree) is measured and recorded.
Performance measurement- Single-leg hop test | 5 months
  Single-leg hop tests are implemented. Right and left hop results are recorded in cm.
Performance measurement- vertical jump tests | 5 months
  Vertical jump tests are implemented. Results are recorded in cm.
Muscle force measurement | 5 months
  The strength of the gastrocnemius medialis, lateralis and soleus muscles is measured and recorded in Newtons.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Gözener Canbülbül, PhD(c), Principal Investigator — İstanbul Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Kavacık, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ward SR, Winters TM, Blemker SS. The architectural design of the gluteal muscle group: implications for movement and rehabilitation. J Orthop Sports Phys Ther. 2010 Feb;40(2):95-102. doi: 10.2519/jospt.2010.3302. PMID 20118527
- [Background] Gans C, Bock WJ. The functional significance of muscle architecture--a theoretical analysis. Ergeb Anat Entwicklungsgesch. 1965;38:115-42. No abstract available. PMID 5319094
- [Background] Gans C, de Vree F. Functional bases of fiber length and angulation in muscle. J Morphol. 1987 Apr;192(1):63-85. doi: 10.1002/jmor.1051920106. PMID 3455200
- [Background] Lieber RL, Friden J. Functional and clinical significance of skeletal muscle architecture. Muscle Nerve. 2000 Nov;23(11):1647-66. doi: 10.1002/1097-4598(200011)23:113.0.co;2-m. PMID 11054744
- [Background] Narici MV, Binzoni T, Hiltbrand E, Fasel J, Terrier F, Cerretelli P. In vivo human gastrocnemius architecture with changing joint angle at rest and during graded isometric contraction. J Physiol. 1996 Oct 1;496 ( Pt 1)(Pt 1):287-97. doi: 10.1113/jphysiol.1996.sp021685. PMID 8910216
- [Background] Fukunaga T, Ichinose Y, Ito M, Kawakami Y, Fukashiro S. Determination of fascicle length and pennation in a contracting human muscle in vivo. J Appl Physiol (1985). 1997 Jan;82(1):354-8. doi: 10.1152/jappl.1997.82.1.354. PMID 9029238
- [Background] Wickiewicz TL, Roy RR, Powell PL, Edgerton VR. Muscle architecture of the human lower limb. Clin Orthop Relat Res. 1983 Oct;(179):275-83. PMID 6617027
- [Background] Kawakami Y, Ichinose Y, Fukunaga T. Architectural and functional features of human triceps surae muscles during contraction. J Appl Physiol (1985). 1998 Aug;85(2):398-404. doi: 10.1152/jappl.1998.85.2.398. PMID 9688711
- [Background] Kwah LK, Pinto RZ, Diong J, Herbert RD. Reliability and validity of ultrasound measurements of muscle fascicle length and pennation in humans: a systematic review. J Appl Physiol (1985). 2013 Mar 15;114(6):761-9. doi: 10.1152/japplphysiol.01430.2011. Epub 2013 Jan 10. PMID 23305989